CLINICAL TRIAL: NCT01684709
Title: Enhancing Informal Caregiving to Support Diabetes Self-Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, James Aikens, PhD, Associate Professor of Family Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DK088294; 1R18DK088294-01 (NIH)
Record Dates: First submitted 2012-08-22; First posted 2012-09-13 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes; Informal Caregivers; Self Care; Quality of Life; Health Information Technology
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telemonitoring + self-management support (Experimental): Automated assessment calls with follow-up by a Care Manager and a CarePartner for 12 months. Baseline, 6 month, and 12 month follow-up.
  Interventions: Behavioral: Telemonitoring + self-management support
- Usual Care (No Intervention): Usual Care

INTERVENTIONS:
Behavioral: Telemonitoring + self-management support — Weekly automated assessment calls with follow-up by a care manager and a CarePartner for 12 months. Baseline, 6 month, and 12 month follow-up
  Arms: Telemonitoring + self-management support

SUMMARY:
This study compares the medical and psychological effects of telemonitoring plus intensified self-management support to those of usual care alone for patients with poorly controlled type 2 diabetes mellitus (DM). If this intervention proves effective without increasing costs or clinician burden, then its implementation could yield major public health benefits, especially for vulnerable and underserved DM patients, and broader societal benefit may occur through increased helping behavior and strengthened social ties.

DETAILED DESCRIPTION:
Although in-home caregivers (ICGs) help improve diabetes mellitus (DM) outcomes, they may lack the resources needed to do this optimally, and are at risk for psychosocial decline and caregiver burnout. Complicating matters, millions of chronically-ill older Americans live alone and receive long-distance caregiving without any supporting structure or resources to ensure its effectiveness. In this study, diabetes patients with poor glycemic will be recruited from two clinical sites, and half will have an ICG. Patients will nominate a "CarePartner" (CP; adult relatives or friends from outside their home) to receive weekly email reports about their DM health and behavioral needs, and will be given resources to help them to provide self-management support. Patients will then be randomized to receive either one year of CP intervention or usual medical care. In the CP intervention arm, patients will provide weekly updates on their DM health and self-management through weekly automated telemonitoring. Summaries of this will be emailed to their CP along with guidance on helping the patient address reported problem(s), and their clinicians will be alerted about medically-urgent problems. We will assess the following outcomes in both arms before intervention and also after 6 and 12 months of intervention: glycemic control, DM-related distress, DM self-management, health-related quality of life, systolic blood pressure, caregiver burden, relationship quality, and cost of DM care.

ELIGIBILITY:
Inclusion criteria:

* type 2 DM (hospitalization or outpatient visit within 12 months for >2 ICD9 codes of 250.xx or therapeutic class codes C4G, C4K, or C4L in past 2 years' problem list)
* poor glycemic control (recent HbA1c% >7.5)
* at least 21 years old
* fluent in English
* can use telephone numeric touchtone keypad
* can identify 1-4 eligible CPs
* not in palliative care, on transplant waitlist, or at high risk for 1-year mortality
* free of major psychiatric or cognitive impairment.
* ICGs: We will stratify recruitment within sites so that 50% of enrolled patients have an ICG.
* Patients with an ICG cannot enroll unless their ICG also provides consent.
* has a CP that resides in continental US but outside patient's household; has communicated with patient, in person or by phone, at least once monthly over preceding 6 months; has a home telephone or mobile cell phone; has an internet connection; can communicate via e-mail; is free of severe psychiatric/cognitive impairment; is fluent in English; and is at least 21 years of age.

Exclusion criteria

* Limited life expectancy (e.g., advanced stage cancer/heart failure/on oxygen/end stage renal disease), receiving palliative care
* active alcohol or drug abuse
* dementia, bipolar disorder, schizophrenia
* unable to speak English
* not planning to get all or most of care at study site
* primary care physician not affiliated with study site
* unable to use a telephone to respond to weekly automated self-management support calls
* unable to nominate an eligible CP
* ICG (if present) does not consent to participate.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 864 (Actual)
Dates: Start 2012-12; Primary Completion 2017-09-26 (Actual); Study Completion 2017-09-26 (Actual)

PRIMARY OUTCOMES:
12-month glycemic control | 12 months
  H1 (Primary biological outcome): Compared to DM patients randomized to control, those randomized to intervention will have a 0.3% greater improvement in HbA1c units.

SECONDARY OUTCOMES:
Secondary effects upon adjustment to diabetes | 12 months
  Compared to controls, intervention patients will have lower diabetes related distress.

CONTACTS AND LOCATIONS:
Overall Officials: James E Aikens, PhD, Principal Investigator — University of Michigan
Locations (6):
- United States (6):
  - University of Michigan, Ann Arbor, Michigan
  - Hamilton Health Center, Flint, Michigan
  - Center for Family Health, Jackson, Michigan
  - Alcona Health Center, Lincoln, Michigan
  - Muskegon Family Care, Muskegon Heights, Michigan
  - St. John Masonic Medical Center, Saint Clair Shores, Michigan

IPD SHARING:
Plan to Share IPD: Undecided
Pending IRB approval.